CLINICAL TRIAL: NCT05609656
Title: Calcium Electroporation in Combination With Irreversible Electroporation and Immunotherapy in Patients With Proficient Mismatch Repair System (pMMR) Metastatic Colorectal Cancer - A Prospective, Phase 2 Study
Brief Title: Electroporation and Immunotherapy in Metastatic Colorectal Cancer
Acronym: ELI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated on the basis on an evaluation of the efficacy and safety of the 4 included and treated patients.
Sponsor: Ismail Gögenur (Other)
Responsible Party: Sponsor-Investigator, Ismail Gögenur, Professor, Zealand University Hospital
Organization: Zealand University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-500045-25-00
Record Dates: First submitted 2022-10-27; First posted 2022-11-08 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Irreversible electroporation; Calcium electroporation; Pembrolizumab; Abscopal effect
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Electroporation; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- IRE + CaEP + Pembrolizumab (Experimental): Irreversible electroporation (IRE) and calcium electroporation (CaEP) on Day 1, followed by Pembrolizumab on Day 2 (+4 days) and then every 3 weeks (q3w) for up to 12 months in total.
  Interventions: Device: Irreversible electroporation; Device: Calcium electroporation; Drug: Pembrolizumab

INTERVENTIONS:
Device: Irreversible electroporation — Percutaneous ablation of a metastatic lesion.
  Irreversible electroporation is delivered through the NanoKnife system (AngioDynamics, New York, USA). The system is CE approved for medical use.
  Other Names: (IRE)
Device: Calcium electroporation — Just before the reversible electroporation, calcium chloride will be injected into the primary tumor. The electroporation will be delivered as at least four pulses and up to eight pulses. The device is repositioned after each pulse to ensure coverage of the entire surface area of the tumor.
  The reversible electroporation regime will be delivered through the endoscopic device EndoVE®, while the ePORE® will be used for pulse generation, both CE approved.
  Other Names: (CaEP)
Drug: Pembrolizumab — Pembrolizumab 200 mg as an IV infusion every 3 weeks (+/- 3 days) for up to 12 months
  Pembrolizumab is an immune checkpoint inhibitor (PD-1-inhibitor).
  Other Names: Keytruda

SUMMARY:
The trial is designed as an investigator initiated prospective phase 2 study in patients with metastatic pMMR colorectal cancer (CRC) to determine the safety and efficacy of calcium electroporation (CaEP) performed concurrently with irreversible electroporation (IRE) followed by a PD-1 inhibitor (pembrolizumab).

DETAILED DESCRIPTION:
The investigators hypothesize that Ca-EP targeting the primary CRC tumor combined with IRE targeting a metastasis will be a promising, safe two target approach to ensure sufficient immune response both locally and systemic to potentiate the efficacy of immunotherapy in patients with pMMR metastatic CRC.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age ≥ 18 years of age
3. Histologically confirmed stage IV, non-resectable pMMR colorectal cancer
4. The primary malignant tumor is left sided (cancer of the splenic flexure and cancer in regions distal to the splenic flexure, including the rectum)
5. The primary tumor is described as reachable at index endoscopy
6. At least two metastatic tumors must be present. One metastatic tumor, that in the opinion of the investigators is amenable to IRE, and at least one additional metastatic tumor that will not undergo IRE. Both lesions must be accessible for biopsy
7. Previous chemotherapy a), or b):

   1. Patients refractory to, intolerable of, or refusing standard chemotherapy options including 5-FU, irinotecan, oxaliplatin, bevacizumab and EGFR-inhibitors e.g. panitumumab/cetuximab (if RAS/RAF wild type)
   2. Patients with favourable biological disease, characterized by

   i. Non-progressive disease ≥ 6 months after last administration of prior 1st line chemotherapy or ≥ 18 months since diagnosis of metastatic disease

1. Patients in this category must have been exposed to an EGFR-inhibitor if RAS/RAF wild type

8. Life expectancy greater than 3 months

9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

10. Adequate bone marrow function:

a. Hemoglobin ≥ 5.6 mmol/L or ≥ 9 g/dL, b. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L c. Platelet count ≥ 75 × 109/L

11. Adequate kidney function:

a. Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min or creatinine ≤1.5 X upper limit of normal (ULN)

12. Adequate liver function:

a. Total bilirubin ≤ 1.5 × ULN b. Alanine aminotransferase (ALT): ≤2.5 X ULN or ≤5 X ULN for subjects with liver metastases c. Aspartate aminotransferase (AST): ≤2.5 X ULN or ≤5 X ULN for subjects with liver metastases d. Albumin: >25 g/L

13. Adequate coagulation function:

a. International Normalized Ratio (INR) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as prothrombin Time (PT) or partial prothrombin time (PTT) is within therapeutic range of intended use of anticoagulants b. Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

14. Follow the conditions regarding fertility, pregnancy, or lactation:

1. Female and male participants of reproductive potential (for definition refer to appendix 16.1) must agree to avoid becoming pregnant or impregnating a partner, respectively, while receiving pembrolizumab and for 120 days after the last dose
2. Participants of reproductive potential must use (or have their partner use) an acceptable method of contraception, as outlined in appendix 16.1, during heterosexual activity, while receiving pembrolizumab and for 120 days after the last dose
3. Women of reproductive potential (WORP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to receiving the first dose of pembrolizumab.
4. Women must not be breastfeeding.

Exclusion Criteria:

1. Prior treatment with an immune checkpoint inhibitor (e.g., anti-PD-1, anti-PD-L1, anti-PD-L2 agent, or anti-CTLA-4 agent)
2. Concurrent treatment with an investigational medicinal product
3. Radiotherapy or major surgery within the last two weeks prior to entering the study
4. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results E.g

   1. Uncorrectable coagulation disorder.
   2. Highly inflamed gastrointestinal tissue which is ulcerated and bleeding
   3. Known history of, or any evidence of interstitial lung disease or active, non-infectious pneumonitis
   4. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
5. Patients should be excluded if they have an active, known or suspected autoimmune disease (except thyroiditis with replacement therapy and type I diabetes mellitus).
6. Patients should be excluded if they have a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies), active chronic, acute hepatitis B (e.g., HBsAg reactive), or hepatitis C (e.g., HCV RNA is detected).
7. Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
8. Allergies and Adverse Drug Reaction:

   i. History of allergy to study drug components ii. History of severe hypersensitivity reaction to any monoclonal antibody
9. Patients are excluded if they have active brain metastases or leptomeningeal metastases. Subjects with brain metastases are eligible if metastases have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for [lowest minimum is four weeks or more] after treatment is complete and within 28 days prior to the first dose of nivolumab administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least two weeks prior to study drug administration
10. Absolute contraindications for IRE:

    1. Implanted pacemaker or ICD unit.
    2. History of epilepsy
    3. History of cardiac (ventricular) arrhythmia
    4. Recent myocardial infarction
    5. Congestive heart failure (>NYHA class 2)
    6. Uncontrollable hypertension
11. Relative contraindications for IRE:

    1. Atrial fibrillation
    2. Combined severe stenosis of the common hepatic artery and main portal vein branch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
The incidence rate of adverse events according to CTCAE v. 4.0 | up to 1 month after end of treatment
  Safety of electroporation and immunotherapy according to CTCAE v. 4.0

SECONDARY OUTCOMES:
Tumor response by CT | Baseline compared to 2, 5, 8, 11 months after start of treatment
  Based on CT chest/abdomen scans according to RECIST version 1.1
Tumor response by ultrasound | Baseline compared to 2 months after start of treatment
  Based on contrast enhanced ultrasound (CEUS) utilizing the standardized and quantitative method Dynamic CEUS (DCEUS)
Progression free survival | From start of treatment until unequivocal disease progression, assessed up to 5 years
Overall survival | From start of treatment until unequivocal disease progression, assessed up to 5 years

OTHER OUTCOMES:
immune infiltration by CD3, CD4, and CD8 staining | Baseline compared to 17 days and 2 months after start of treatment
  immune-related treatment-induced changes
immune infiltration by PD-1 and PD-L1 staining | Baseline compared to 17 days and 2 months after start of treatment
  immune-related treatment-induced changes

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No